CLINICAL TRIAL: NCT07271082
Title: Efficacy and Safety of Home-based Structured Physical Exercise in Patients With Acute Ischemic Stroke: a Randomized Controlled, Open-label, Blinded Endpoint Trial-2 (HOPE-STROKE 2)
Brief Title: Efficacy and Safety of Home-based Structured Physical Exercise in Patients With Acute Ischemic Stroke
Acronym: HOPE-STROKE 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOPE-STROKE 2
Record Dates: First submitted 2025-11-27; First posted 2025-12-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Physical Exercise
MeSH Terms: conditions — Ischemic Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (Experimental): Home-based structured physical exercise guidance.
  Interventions: Behavioral: Exercise intervention
- Control group (No Intervention): Subjects will not receive structured physical exercise guidance but are encouraged to engage in regular physical exercise.

INTERVENTIONS:
Behavioral: Exercise intervention — Subjects will undergo 90 days of home-based structured physical exercise guidance.
  Arms: Exercise intervention group

SUMMARY:
This study is a randomized controlled, open-label, blinded endpoint trial. The investigators aim to assess the efficacy and safety of home-based structured physical exercise in participants with acute ischemic stroke.

DETAILED DESCRIPTION:
The study population is participants with acute ischemic stroke within 14 days of onset. All participants are randomly assigned to the exercise intervention group or the control group in a 1:1 ratio. In the exercise intervention group, participants will undergo 90 days of home-based structured physical exercise guidance. The individualized exercise prescription will be determined based on each participant's overall condition. In the control group, participants will not receive structured physical exercise guidance but are encouraged to engage in regular physical exercise. Both groups of participants will receive standard medical management based on the latest guidelines from the American Heart Association/American Stroke Association.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater, male or female;
2. Acute ischemic stroke onset within 14 days;
3. modified Rankin scale (mRS) score ≤ 3;
4. Signed informed consent from the patients or the legally authorized representatives.

Exclusion Criteria:

1. Stroke progression within the past 3 days (defined as an increase in NIHSS score of ≥4 points or an increase in any single item of ≥2 points);
2. Concurrent osteoarthritis, fractures, deep vein thrombosis, unstable angina, severe heart diseases, respiratory diseases, or amputation that may theoretically make it difficult for participants to complete the physical exercise or ambulation;
3. Concurrent movement disorders such as Parkinson's disease or Parkinsonism;
4. Patients who have engaged in regular aerobic physical activity within the past 6 months, defined as more than 150 minutes of moderate-intensity aerobic physical activity; or more than 75 minutes of vigorous-intensity aerobic physical activity; or an equivalent combination of moderate- and vigorous-intensity activity throughout the week;
5. Unable to comply with the study procedures or follow-up due to psychiatric, cognitive, or emotional disorders;
6. Known pregnancy or lactation, or a positive pregnancy test;
7. Currently participating in another drug or device study;
8. Life expectancy less than 1 year;
9. Unable to communicate using a smartphone;
10. Other conditions considered by investigators to be unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Test Distance | Between baseline and 90 days

SECONDARY OUTCOMES:
Proportion of patients with mRS score 0-1 | 90 days
  The mRS ranges from 0 to 6, with higher scores indicating worse outcomes.
Physical Activity Scale for the Elderly (PASE) score | 90 days
  This test assesses physical activity, including leisure, household, and occupational activity. Score range: minimum 0 to maximum 400 or more. Higher score means a better outcome.
Short Physical Performance Battery (SPPB) score | 90 days
  This test measures levels of lower extremity function. The SPPB ranges from 0 to 12, with higher scores indicating better outcomes.
Mean daily step count | 90 days
Patient Health Questionnaire-9 (PHQ-9) score | 90 days
  This test screens for depression. The PHQ-9 ranges from 0 to 27, with higher scores indicating worse outcomes.
Mini Montreal Cognitive Assessment score | 90 days
  This test measures levels of cognitive function. This test ranges from 0 to 15, with higher scores indicating better outcomes.
Resting heart rate | 90 days
Resting blood pressure | 90 days
EQ-5D-5L and EQ-VAS | 90 days
  The EQ-5D-5L includes 5 dimensions: mobility, self-care, usual activities,pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicate worse quality of life.

OTHER OUTCOMES:
Rate of Falls | Within 90 days after randomization
All-cause death | Within 90 days after randomization

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Taihe Hospital of Traditional Chinese Medicine, Fuyang, Anhui
  - Suzhou Municipal Hospital, Suzhou, Anhui
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Xihua County People's Hospital, Zhoukou, Henan
  - Shihezi People's Hospital, Shihezi, Xinjiang
  - Xuanwu Hospital, Capital Medical University, 100053, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Related data will be shared if full study protocol and statistical analysis plan are provided with reasonable design.